CLINICAL TRIAL: NCT02322489
Title: Efficacy of Microcurrent Therapy After Eccentric Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Christophe Demoulin, Main investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Microcurrent
Record Dates: First submitted 2014-12-06; First posted 2014-12-23 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: microcurent; pain; flexibility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham microcurrent therapy (Sham Comparator): The participant is lying on an examination table for one hour; several electrodes are placed over the muscles involved in the provocative task. The microcurrent therapy is then started but it lasts only for 5 seconds.
  Interventions: Device: Sham microcurrent therapy
- Microcurrent Group (Experimental): The participant is lying on an examination table for one hour; several electrodes are placed over the muscles involved in the provocative task. The microcurrent therapy is then started.
  Interventions: Device: Microcurrent Therapy

INTERVENTIONS:
Device: Microcurrent Therapy — Several electrodes are placed over the muscles involved in the provocative task. The microcurrent therapy is then started and lasts for one hour.
  Arms: Microcurrent Group
Device: Sham microcurrent therapy — Several electrodes are placed over the muscles involved in the provocative task. The microcurrent therapy is then started but lasts only for five seconds.
  Arms: Sham microcurrent therapy

SUMMARY:
15 participants will be included in the present study. They will attend two groups of three sessions (i.e. sessions 1-2-3 and sessions 4-5-6) spaced by 3 months:

* session 1 and 4 (performed a few days before the experimental session): session for participants to get familiarized with the test battery.
* session 2 and 5: experimental session (the test battery followed by the provocative task, the test battery, the one-hour "treatment" and the test battery again).
* session 3 and 6 (performed 2 days later): the test battery.

The test battery included flexibility, functional, pressure pain threshold tests.

The provocative task was an isokinetic eccentric task for knee flexors and extensors.

The treatment was either a microcurrent therapy or a placebo microcurrent therapy.

DETAILED DESCRIPTION:
Objective:

To study the efficacy of microcurrent to reduce DOMS (Delayed Onset Muscle Soreness) occuring after an eccentric exercise

Methods:

Experimental protocol

Participants will attend two groups of three sessions (i.e. sessions 1-2-3 and sessions 4-5-6) spaced by 3 months:

* session 1 and 4 (performed a few days before the experimental session): session for participants to get familiarized with the test battery.
* session 2 and 5: experimental session: the test battery followed by the provocative task, the test battery, the one-hour "treatment" (real microcurrents at one of the session and placebo microcurrents at the other one) and the test battery again.
* session 3 and 6 (performed 2 days later): the test battery.

Before starting session 2, patients will be randomized into the microcurrent group or the placebo microcurrent group. Three months later, participants will change of group.

The Test Battery: it will be conducted by a blind (to the treatment) investigator. It will include knee flexor and extensor flexibility tests, a functional test (unilateral " counter-movement jump "), a pain to measure pain threshold of thigh muscles and an isometric maximal voluntary contraction (MVC) test of knee flexors and extensors.

The Provocative task: 40 isokinetic eccentric contractions of knee flexors and extensors.

The one-hour Treatment: with the participant lying on an examination table, several electrodes were located over the muscles involved in the provocative task. The microcurrent therapy was then started. It was stopped after 5 seconds in the "Placebo group" and after one hour in the real "Microcurrent group". The microcurrents were delivered by the machine B-E-St®.

Follow-up: in addition to the 48hours follow-up (session 3/6), participants will fill in a pain visual analogue scale each day after the session 2/5.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic subjects

Exclusion Criteria:

* practice of sports >3h per week
* present pain in the lower limbs
* history of thigh muscle injuries
* recent injury (last 3 months) of the lower limbs
* recent (last 3 months) plyometric exercises or lower limbs strengthening program.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Intensity of pain (Visual analogue scale) | baseline, post-provocative task, post-treatment, 48h follow-up, following days until pain disappears

SECONDARY OUTCOMES:
Flexibility of quadriceps and hamstrings muscles | baseline, post-provocative task, post-treatment, 48h follow-up
  Flexibility of quadriceps muscle was assessed by means of the Prone Quadriceps Flexibility test.
  Flexibility of hamstrings was assessed by means of the Straight Leg Raising (SLR) test
Functional test (Unilateral counter-movement jump) | baseline, post-provocative task, post-treatment, 48h follow-up
  Unilateral counter-movement jump
Pain sensibility threshold (Determined by using a dolorimeter) | baseline, post-provocative task, post-treatment, 48h follow-up
  Determined by using a dolorimeter
Isometric strength (Maximal voluntary contraction of knee flexor and extensor muscles) | baseline, post-provocative task, post-treatment, 48h follow-up
  Maximal voluntary contraction of knee flexor and extensor muscles

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Demoulin, PhD, Principal Investigator — University of Liege
Locations (1):
- Liege University Hospital Center, Liège, Liege, Belgium